CLINICAL TRIAL: NCT01847092
Title: An Exploratory Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Design Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AZD1722 in CKD Patients With Type 2 Diabetes Mellitus and Albuminuria
Brief Title: A Study in CKD Patients With Type 2 Diabetes Mellitus and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5610C00001
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
Keywords: albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Albuminuria | interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1722 (Active Comparator): AZD1722 in 5, 15, 30, or 60 mg capsules. Starting dose is 15 mg BID PO for 12 Weeks
  Interventions: Drug: AZD1722
- Placebo (Placebo Comparator): Placebo capsule BID PO for 12 Weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1722
  Arms: AZD1722
Drug: Placebo — Placebo for AZD1722
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the study drug is safe, tolerable and active in reducing albuminuria in patients with Chronic Kidney Disease with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 80 years, inclusive.
* Body mass index between 18 and 45 kg/m2, inclusive.
* Type 2 diabetes mellitus and receiving ≥1 glucose lowering medication for at least 3 months prior to randomization
* Stage 3 CKD
* MSSBP ≥130 mmHg
* Urinary albumin: mean UACR ≥ 200 mg/g

Exclusion Criteria:

* Urinary albumin: UACR > 3500 mg/g
* History of a renal transplant
* MSSBP >180 mmHg or a MSDBP of >120 mmHg on two occasions during screening or run-in periods
* History of inflammatory bowel disease or diarrhea predominant irritable bowel syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Creekside Endocrine Associates PC, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD1722: AZD1722 in 5, 15, 30, or 60 mg capsules. Starting dose is 15 mg BID PO for 12 Weeks
  AZD1722
Period: Overall Study
Arm/Group | AZD1722 | Placebo
Started | 77 | 77
Completed | 51 | 66
Not Completed | 26 | 11
Not completed — Adverse Event | 12 | 3
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Protocol Specified | 8 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1722 | Placebo | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.79) | 65.6 (8.77) | 65.1 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 37
  Not Hispanic or Latino | 59 | 58 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 18 | 39
  White | 53 | 53 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Urine Albumin to Creatinine Ratio (UACR)
Description: The difference between tenapanor and placebo in the change in UACR from baseline to the end of 12 weeks of treatment
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | AZD1722 | Placebo
Number analyzed (Participants) | 77 | 77
mg/g | -64.6 (898.4) | 104.8 (668.0)
Statistical Analysis 1: Comparison: AZD1722 vs Placebo; Test type: Superiority; p = 0.279, Mixed Models Analysis

2. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (mL/Min/1.73 m2) From Baseline to Week 12 Endpoint
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | AZD1722 | Placebo
Number analyzed (Participants) | 77 | 77
mL/min/1.73 m2 | -2.8 (1.21) | -2.7 (1.19)
Statistical Analysis 1: Comparison: AZD1722; Test type: Superiority; p = 0.94, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | AZD1722 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 3/77 | 2/77
Other Adverse Events (participants affected / at risk) | 45/77 | 4/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1722 (N=77) | Placebo (N=77)
Hyperkalemia (Investigations) | 2 (2) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1722 (N=77) | Placebo (N=77)
Diarrhea (Gastrointestinal disorders) | 45 (45) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days